CLINICAL TRIAL: NCT01236326
Title: A Randomized, Prospective, Parallel Group Study of Conventional Laparoscopic Donor Nephrectomy (LDN) Versus Laparoendoscopic Single Site Donor Nephrectomy (LESS-DN) in Living Donor Kidney Transplantation
Brief Title: Conventional Laparoscopic Versus Laparoendoscopic Single Site Donor Nephrectomy in Living Donor Kidney Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1009011249
Record Dates: First submitted 2010-11-04; First posted 2010-11-08 (Estimated); Results first posted 2015-08-26 (Estimated); Last update posted 2019-06-12 (Actual); Status verified 2019-05

CONDITIONS: Living Donors; Nephrectomy; Kidney Transplantation; Surgery, Laparoscopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LESS-DN (Active Comparator)
  Interventions: Procedure: Laparoendoscopic single site donor nephrectomy
- Conventional LDN (Active Comparator)
  Interventions: Procedure: Conventional laparoscopic donor nephrectomy

INTERVENTIONS:
Procedure: Laparoendoscopic single site donor nephrectomy — Patients randomized to this arm will undergo laparoendoscopic single site donor nephrectomy
  Arms: LESS-DN
Procedure: Conventional laparoscopic donor nephrectomy — Patients randomized to this arm will undergo conventional laparoscopic donor nephrectomy
  Arms: Conventional LDN

SUMMARY:
Laparoscopic nephrectomy (removal of the kidney) is the most common procedure for people donating a kidney to be used for living donor kidney transplantation. Laparoscopic donor nephrectomy (LDN) was a great advance in the field of living donor kidney transplantation due to the many advantages it offers over open nephrectomy, including significantly shorter hospitalization and recovery time, and significantly improved cosmetic result related to the nephrectomy scar(s). More recently, a new procedure has been introduced to the field of laparoscopic nephrectomy, called laparoendoscopic single site donor nephrectomy (LESS-DN). In the LESS-DN procedure, a single natural orifice (the umbilicus or belly button) is used as the single incision site through which the entire donor nephrectomy is performed. The LESS-DN procedure may further decrease donor morbidity by further decreasing length of stay, lessening recovery time, and improving satisfaction with the surgical scar. The investigators propose to evaluate conventional LDN versus a LESS-DN in a randomized, controlled trial in living kidney donors. The investigators will compare operative times and intra-operative donor management, intra- and post-operative complications, pain scores, analgesic requirements, length of stay, recovery parameters, surgical scar satisfaction, and function and survival of the transplanted kidney for the two groups of subjects: (1) the group that has the conventional laparoscopic donor nephrectomy; and, (2) the group that has the laparoendoscopic single site donor nephrectomy.

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled to undergo laparoscopic living donor nephrectomy will be eligible for the study.

Exclusion Criteria:

* There are no exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2010-11; Primary Completion 2013-06 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph J Del Pizzo, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- NewYork-Presbyterian Hospital/Weill Cornell Medical Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LESS-DN | Conventional LDN
Started | 50 | 55
Completed | 49 | 51
Not Completed | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LESS-DN | Conventional LDN | Total
Number analyzed (Participants) | 49 | 51 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.8 (11.9) | 47.4 (11.5) | 47.1 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 29 | 58
  Male | 20 | 22 | 42
Race/Ethnicity, Customized [Number; unit: participants]
  African American | 5 | 9 | 14
  Caucasian | 28 | 31 | 59
  Hispanic | 10 | 9 | 19
  All Other | 6 | 2 | 8
Region of Enrollment [Number; unit: participants]
  United States | 49 | 51 | 100
Relationship to Recipient [Number; unit: participants]
  Living Related | 21 | 24 | 45
  Living Unrelated | 28 | 27 | 55
Side of Donation (left) [Number; unit: participants]
  Left | 45 | 48 | 93
  Right | 4 | 3 | 7
Body Mass Index (BMI) [Number; unit: participants]
  BMI < 30 kg/m^2 | 36 | 36 | 72
  BMI >= 30 kg/m^2 | 13 | 15 | 28
Multiple Arteries [Number; unit: participants]
  Yes | 6 | 6 | 12
  No | 43 | 45 | 88

OUTCOME MEASURES:

1. Primary Outcome: The Primary End Point of the Study Was the Mean/Median Number of Days Postsurgery Required for Each Group to Return to 100% Functioning Capacity.
Description: The Primary Endpoint of the Study Will be Patient Self-reported "Return to 100%", as Measured by the Number of Days Post-surgery That the Patient Reports His or Her Return to 100% Functioning Capacity.
Time Frame: 1 year
Population: The number of participants analyzed is lower than the number of baseline participants because overall, 25% of subjects did not return the 2-month questionnaire (26.5% of the LESS-DN group and 23.5% of the Conventional LDN group).
Measure: Mean (Standard Deviation); unit: days
Arm/Group | LESS-DN | Conventional LDN
Number analyzed (Participants) | 36 | 39
days | 43 (15) | 45 (22)

2. Secondary Outcome: Days on Oral Pain Medication After Discharge
Time Frame: 2 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | LESS-DN | Conventional LDN
Number analyzed (Participants) | 36 | 39
days | 6 (4) | 7 (8)

3. Secondary Outcome: Days Before Going Back to Work
Time Frame: 2 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | LESS-DN | Conventional LDN
Number analyzed (Participants) | 36 | 39
days | 24 (14) | 27 (18)

4. Secondary Outcome: Days to Normal Day-to-day Activities
Time Frame: 2 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | LESS-DN | Conventional LDN
Number analyzed (Participants) | 36 | 39
days | 30 (17) | 33 (25)

5. Secondary Outcome: Recovered by 2 Months After Donation
Time Frame: 2 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | LESS-DN | Conventional LDN
Number analyzed (Participants) | 36 | 39
participants | 35 | 31

ADVERSE EVENTS:
Arm/Group | LESS-DN | Conventional LDN
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/51
Other Adverse Events (participants affected / at risk) | 9/49 | 7/51
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LESS-DN (N=49) | Conventional LDN (N=51)
Conversion to Hand Assist Laparoscopy (Renal and urinary disorders) | 3 (3) | 2 (2) — For bleeding, difficult dissection, or difficult mobilization
Ileus within 30 days (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Superficial Surgical Site Infection (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Re-admission (General disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
Inability to secure complete data on the donor questionnaires (25% of subjects did not return 2-month questionnaire); no validated tool available to assess donor recovery and satisfaction; clinical donor follow-up was suboptimal.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes